CLINICAL TRIAL: NCT04438616
Title: Comparison of Patient Satisfaction and Primary Implant Stability Between Two Different Magnetic Attachment for Implant Retained Mandibular Over Denture Following Immediate Loading
Brief Title: Comparison of Patient Satisfaction and Primary Implant Stability Between Two Different Magnetic Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hussein Hatam Jawad, Main-Supervisor :Dr.Ahmed fahmy (Ass.professor of prosthodontics, faculity of dentistry ,cairo university ) \co-supervisor :Amr ahmednaguib (lecturer of prosthodontic ) \ Principle Investigator.:Hussein hatam jawad, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3042020
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-04

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dome magnetic attachment (Active Comparator): * A crestal incision is made using No. 15 c blade extending over the crest of anterior mandible and a full mucoperiosteum flaps elevated to provide access to the alveolar ridge for implant installed.
  * Full sequential drilling under copious saline irrigation will be made as indicated by the company guide lines. insertion of two implant in each group by the contra angle handpiece with special adaptor
  * We connect magnetic attachment(dome) for each groups on complete denture by pick up procedure at day of implant installation
  Interventions: Procedure: dome magnetic attachment
- flat magnetic attachment (Active Comparator): * A crestal incision is made using No. 15 c blade extending over the crest of anterior mandible and a full mucoperiosteum flaps elevated to provide access to the alveolar ridge for implant installed.
  * Full sequential drilling under copious saline irrigation will be made as indicated by the company guide lines. insertion of two implant in each group by the contra angle handpiece with special adaptor
  * We connect magnetic attachment(flat) for each groups on complete denture by pick up procedure at day of implant installation
  Interventions: Procedure: flat magnetic attachment

INTERVENTIONS:
Procedure: dome magnetic attachment — * All patients will receive complete denture before implant installation .
  * The CBCT examination should be take
  * patients received infiltration local anesthesia
  * A crestal incision is made using No. 15 c blade .
  * Full sequential drilling under copious saline irrigation will be made . insertion of two implant by the contra angle handpiece with special adaptor
  * We connect magnetic attachment(dome) on complete denture by pick up procedure at day of implant installation.
  * Implant stability will be measured using smart peg /osstell at the day of implant installation and after 2,4,8,12 weeks.
  * Patient satisfaction measure
  Arms: dome magnetic attachment
Procedure: flat magnetic attachment — * All patients will receive complete denture before implant installation .
  * The CBCT examination should be take
  * patients received infiltration local anesthesia.
  * A crestal incision is made using No. 15 c blade
  * Full sequential drilling under copious saline irrigation will be made as indicated by the company guide lines. insertion of two implant by the contra angle handpiece with special adaptor
  * We connect magnetic attachment(flat) on complete denture by pick up procedure at day of implant installation.
  * Implant stability will be measured using smart peg /osstell at the day of implant installation and after 2,4,8,12 weeks.
  * Patient satisfaction measure in 2 weak and after 12 weak by Denture satisfaction questionnaire
  Arms: flat magnetic attachment

SUMMARY:
* Patients were randomly divided in to two groups by using computerized software ; the first group received flat magnetic attachment design while the second group received dome magnetic attachment design.which the inclusion criteria is completely edentulous patient ,Age range from 40 to 70 year old ,skeletal class 1, both sexes
* Implant stability will be measured for both groups using smart peg /osstell at the day of implant installation and after 2,4,8,12 weeks.
* Patient satisfaction measure in 2 weak and after 12 weak by Denture satisfaction questionnaire

DETAILED DESCRIPTION:
* The selected patients will be informed of the nature of the research work and informed consent will be obtained then randomized in equal proportions between control group flat magnetic attachment design and study group dome magnetic attachment design technique
* Radiographic examination included a preoperative digital panoramic radiograph with 1:1 magnification for each patient as a primary survey to obtain an approximation of the available bone height and detect the presence of remaining roots and localized pathosis.
* All patients will receive complete denture before implant installation .Constructed as the following
* Primary impression to construct diagnostic cast and special tray .
* Secondary impression with selective pressure impression technique to have master caste and occlusion block
* Face bow transfer and centric relation record will be utilized to mount the master cast on semi adjuctable articulator ,then setting the teeth and trying the denture in patient mouth.
* Processing of acrylic and lab remounting ,then delivery of the denture.
* The complete denture will be duplication to be used as a guide to fabricate the radiographic stent after placement radio opaque marker in two lower canines then send patient to perform CBCT and these duplicate denture use as surgical template to place two implant.
* CBCT machine: planmeca / CBCT soft ware : blue sky / FOV: single arch mandible /voxel size :400 Mm ( KV:90 / MA: 8 / S:11,997)
* The CBCT examination where performed in radiology department / collage of dentistry /cairo university
* serial follow up CBCT not need
* Patients were randomly divided in to two groups by using computerized software ; the first group received flat magnetic attachment design while the second group received dome magnetic attachment design e. All surgeries were performed by the same prosthodontic.
* All surgical procedures were performed under strict aseptic conditions, all patients received infiltration local anesthesia (Articaine 4% 1:100 000 epinephrine).
* A crestal incision is made using No. 15 c blade extending over the crest of anterior mandible and a full mucoperiosteum flaps elevated to provide access to the alveolar ridge for implant installed.
* Full sequential drilling under copious saline irrigation will be made as indicated by the company guide lines. insertion of two implant in each group by the contra angle handpiece with special adaptor.(control and study groups)
* The flap will then be closed using interrupted 4/0 resorbable sutures.
* We connect magnetic attachment(flat,dome) for each groups on complete denture by pick up procedure at day of implant installation.
* Relief space from the denture for the magnetic attachment will be made and a rubber dam will be used to closed the under cute under the magnetic attachment. pickup material will be added in the relief area to connect the housing to the denture intra orally.
* Implant stability will be measured for both groups using smart peg /osstell at the day of implant installation and after 2,4,8,12 weeks.
* Patient satisfaction measure in 2 weak and after 12 weak by Denture satisfaction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patient.
* Age range from 40 to 70 year old
* Skeletal class 1
* Both sexes.

Exclusion Criteria:

* No intra oral soft and hard tissue pathology
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Patient with sever parafunctional occlusal activity.
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability,.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
name of measurement: Patient satisfaction | Patient satisfaction measure in 2 weak
  Denture satisfaction questionnaire
name of measurement: Patient satisfaction | Patient satisfaction measure in 12 weak
  Denture satisfaction questionnaire

SECONDARY OUTCOMES:
name of measurement: implant stability | Implant stability will be measure at day of implant
  Measurement unit: ISQ \ Measurement device: Osstell device \ scale: 1-100 ISQ .measurement tool is smart peg attached to implant and hand-held probe.
name of measurement: implant stability | Implant stability will be measure after 2 weak
  Measurement unit: ISQ \ Measurement device: Osstell device \ scale: 1-100 ISQ .measurement tool is smart peg attached to implant and hand-held probe.
name of measurement: implant stability | Implant stability will be measure after 4 weak
  Measurement unit: ISQ \ Measurement device: Osstell device \ scale: 1-100 ISQ measurement tool is smart peg attached to implant and hand-held probe.
name of measurement: implant stability | Implant stability will be measure after 8 weak
  Measurement unit: ISQ \ Measurement device: Osstell device \ scale: 1-100 ISQ measurement tool is smart peg attached to implant and hand-held probe.
name of measurement: implant stability | Implant stability will be measure after 12 weak
  Measurement unit: ISQ \ Measurement device: Osstell device \ scale: 1-100 ISQ measurement tool is smart peg attached to implant and hand-held probe.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Boerrigter EM, Geertman ME, Van Oort RP, Bouma J, Raghoebar GM, van Waas MA, van't Hof MA, Boering G, Kalk W. Patient satisfaction with implant-retained mandibular overdentures. A comparison with new complete dentures not retained by implants--a multicentre randomized clinical trial. Br J Oral Maxillofac Surg. 1995 Oct;33(5):282-8. doi: 10.1016/0266-4356(95)90038-1. PMID 8555143
- [Background] Allen PF, McMillan AS, Walshaw D. A patient-based assessment of implant-stabilized and conventional complete dentures. J Prosthet Dent. 2001 Feb;85(2):141-7. doi: 10.1067/mpr.2001.113214. PMID 11208203
- [Background] Feine JS, Carlsson GE, Awad MA, Chehade A, Duncan WJ, Gizani S, Head T, Lund JP, MacEntee M, Mericske-Stern R, Mojon P, Morais J, Naert I, Payne AG, Penrod J, Stoker GT, Tawse-Smith A, Taylor TD, Thomason JM, Thomson WM, Wismeijer D. The McGill consensus statement on overdentures. Mandibular two-implant overdentures as first choice standard of care for edentulous patients. Montreal, Quebec, May 24-25, 2002. Int J Oral Maxillofac Implants. 2002 Jul-Aug;17(4):601-2. No abstract available. PMID 12182304
- [Background] Tallgren A. The continuing reduction of the residual alveolar ridges in complete denture wearers: a mixed-longitudinal study covering 25 years. J Prosthet Dent. 1972 Feb;27(2):120-32. doi: 10.1016/0022-3913(72)90188-6. No abstract available. PMID 4500507
- [Background] Barao VA, Assuncao WG, Tabata LF, Delben JA, Gomes EA, de Sousa EA, Rocha EP. Finite element analysis to compare complete denture and implant-retained overdentures with different attachment systems. J Craniofac Surg. 2009 Jul;20(4):1066-71. doi: 10.1097/SCS.0b013e3181abb395. PMID 19553853